CLINICAL TRIAL: NCT02398292
Title: Meals, Mindfulness & Moving Forward: A Multi-modal Approach to Addressing Cardiovascular Risk and Building Resilience in Youth Suffering From Psychosis
Brief Title: A Multi-modal Approach to Addressing Cardiovascular Risk and Building Resilience in Youths With Psychosis
Acronym: M3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Lynne Shinto, Associate Professor, Oregon Health and Science University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10376
Record Dates: First submitted 2015-03-20; First posted 2015-03-25 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Schizophrenia; Psychotic Disorders
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Meals; Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- M3 Program (Other): Non-randomized experimental group. The program is a six-week multi-modal intervention, including nutrition education and cooking classes, physical activity, and mindfulness. Outcomes will be compared to a non-randomized control group.
  Interventions: Other: M3 Program
- Control (Other): Non-randomized control group. Outcomes will be compared at same time points (baseline, 6 weeks, 12 weeks).
  Interventions: Other: Control

INTERVENTIONS:
Other: M3 Program — Participants and their study partners will learn about food, movement, and mindfulness through hands-on curriculum.
  Other Names: Meals, Mindfulness and Moving Foward Program
  Arms: M3 Program
Other: Control — Participants will not participate in M3 program but will have same outcomes measured at same time points (baseline, 6 weeks, 12 weeks).
  Arms: Control

SUMMARY:
The purpose of this study is to determine the feasibility (≥ 50% completion rate) of a 6-week nutrition, movement, and mindfulness program for youth with recent diagnosis of psychosis.

DETAILED DESCRIPTION:
The purpose of this study is to determine the feasibility of a 6-week nutrition, movement, and mindfulness program (M³ Program) for youth with a recent diagnosis of psychosis. Program effects on metabolic and mental health outcomes compared to wait-list control will also be assessed. Participants will be 15-25 years of age, and have a recent diagnosis of psychosis. Twenty participants and their study partners (20 study partners) will be equally divided into two cohorts. Participants will sign up for one of the two series on a rolling enrollment basis until both of the program date frames are filled. Participants that signed up for the second series will serve as a wait-list control; outcomes from the participants in the first series will be compared to this group. M³ will be a combination of didactic and experiential training. The course will meet once-a-week for six weeks. Participants will learn how to prepare healthy snacks and meals, make healthy choices when eating out, and interpret food packaging and labels. They will also learn about different forms of mindfulness exercises and movement, such as yoga, martial arts, and a Japanese style of drumming. Feasibility will be assessed throughout the program.

ELIGIBILITY:
Inclusion Criteria:

* First diagnosis of psychosis occurs within 3 years of enrollment into the study or are a graduate of the Early Assessment and Support Alliance Program (EASA).
* Established mental health provider and primary care physician.
* Age 15 to 25 years (inclusive)
* Able to enroll with a study partner (study partner can be a healthy volunteer)
* Able to read and write in English

Exclusion Criteria:

* Active suicidal or homicidal thoughts
* Mental status exam which suggests high risk for disruptiveness to group process or danger to self and others.
* If a graduate of EASA, the participant must have a primary care or mental health provider.

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2015-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Feasibility assessed by 6-week program completion by 50% of participants attending at least 60% of the program | 6 weeks

SECONDARY OUTCOMES:
Body Mass Index | 6 and12 weeks
  body mass index
Waist Circumference | 6 and12 weeks
  waist circumference measured in cm
Lipid Panel | 6 and12 weeks
  total cholesterol, triglycerides, HDL, LDL
Quick Scale for the Assessment of Negative Symptoms and Positive Symptoms | 6 and12 weeks
  A rating scale to measure positive symptoms of schizophrenia. The QSANS-QSAPS assessment is administered by a trained health professional and takes 30 to 45 minutes to complete.
Connor-Davidson Resilience Scale | 6 and12 weeks
  A measurement of 'hardiness', or one's ability to successfully cope with stress. The scale draws on a number of resilient characteristics, including patience, tolerance to negative affect, sense of humor, commitment, recognition of limits to control, engaging the support of others, and adaptability. The CD-RISC contains 25 items and asks subjects to rate how they felt over the past month on a Likert-type scale. Total score range is 0 - 100, with higher scores indicating higher levels of resiliency.
Quality of LIfe - SF12 | 6 and12 weeks
  : The SF-12 is a 12-item validated shortened version of the SF-36 and was designed to provide a health related quality of life measure that was quick and easy to administer in large population studies. The SF-12 contains a subset of the 12 items from the SF-36 and information from this subset of questions is used to construct a physical and mental component summary score.

CONTACTS AND LOCATIONS:
Overall Officials: Lynne Shinto, ND, MPH, Principal Investigator — Oregon Health and Science University; Craigan Usher, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No